CLINICAL TRIAL: NCT05878860
Title: A Phase 1/2, Open-Label, Dose Escalation and Dose Expansion Study to Evaluate the Safety and Tolerability of ATSN-201 Gene Therapy in Male Subjects With RS1-Associated X-linked Retinoschisis
Brief Title: ATSN-201 Gene Therapy in RS1-Associated X-linked Retinoschisis
Acronym: LIGHTHOUSE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Atsena Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ATSN-201-1
Record Dates: First submitted 2023-05-12; First posted 2023-05-26 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: X-linked Retinoschisis
Keywords: XLRS, RS1
MeSH Terms: conditions — Retinoschisis

STUDY DESIGN:
Masking Description: Cohort 3 will be partially masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort 1, Low Dose (Experimental)
  Interventions: Biological: ATSN-201
- Cohort 2, High Dose (Experimental)
  Interventions: Biological: ATSN-201
- Cohort 3, Mid Dose (Experimental)
  Interventions: Biological: ATSN-201
- Cohort 4, Low Volume (Experimental)
  Interventions: Biological: ATSN-201
- Cohort 4, High Volume (Experimental)
  Interventions: Biological: ATSN-201
- Cohort 4, Control (No Intervention)
- Cohort 5, Pediatric (Experimental)
  Interventions: Biological: ATSN-201

INTERVENTIONS:
Biological: ATSN-201 — AAV.SPR-hGRK1-hRS1syn
  Arms: Cohort 1, Low Dose; Cohort 2, High Dose; Cohort 3, Mid Dose; Cohort 4, High Volume; Cohort 4, Low Volume; Cohort 5, Pediatric

SUMMARY:
This study will evaluate the safety and tolerability of ATSN-201 in male subjects ≥ 6 years of age with RS1-associated X-linked retinoschisis (XLRS).

DETAILED DESCRIPTION:
Eligible patients who enroll in this study will receive a one-time subretinal injection of ATSN-201 in one eye. Safety and tolerability will be evaluated for 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 for Cohorts 1 through 3, and age ≥ 6 years and < 18 years for Cohort 4.
2. Male patients with clinical diagnosis of XLRS caused by mutations in RS1.
3. Best corrected visual acuity (BCVA) in study eye of 34 to 73 Early Treatment Diabetic Retinopathy Study (ETDRS) letters (corresponding to a Snellen acuity of 20/200 to 20/40).

Exclusion Criteria:

1. Pre-existing eye conditions in the study eye that would contribute significantly to an increased risk of visual loss from a subretinal injection.
2. Any intraocular surgery (including laser treatment) in the study eye within 6 months prior or any intraocular surgery anticipated in the study eye during the first 12 months of the study.
3. Treatment in a prior ocular gene or cell therapy study.

Min Age: 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2023-08-22 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability as assessed by dose-limiting toxicities and treatment-emergent adverse events | From baseline to week 52
  Incidence of dose-limiting toxicities (DLTs) and treatment-emergent adverse events (TEAEs).

SECONDARY OUTCOMES:
Visual acuity as assessed by best-corrected visual acuity | From baseline to week 52
  Change in best-corrected visual acuity (BCVA).
Visual acuity as assessed by low-luminance visual acuity | From baseline to week 52
  Change in low-luminance visual acuity (LLVA).
Visual function as assessed by contrast sensitivity | From baseline to week 52
  Change in contrast sensitivity.
Visual function as assessed by full-field electroretinogram parameters | From baseline to week 52
  Change in full-field electroretinogram (ffERG) parameters.
Visual function as assessed by microperimetry | From baseline to week 52
  Change in microperimetry.
Visual function as assessed by static perimetry | From baseline to week 52
  Change in static perimetry.
Macular structure as assessed by spectral domain optical coherence tomography | From baseline to week 52
  Change in spectral domain optical coherence tomography (SD-OCT).
Macular structure as assessed by fundus autofluorescence | From baseline to week 52
  Change in fundus autofluorescence (FAF).
Subject-reported visual function as assessed by the NEI VFQ-25 in adult subjects | From baseline to week 52
  Change in the National Eye Institute's Visual Function Questionnaire 25 (NEI VFQ-25) score for adult subjects with scores from 0 to 100 where a higher score indicates a better outcome.
Subject-reported visual function as assessed by the CVAQC in pediatric subjects | From baseline to week 52
  Change in the Cardiff Visual Ability Questionnaire for Children (CVAQC) score for pediatric subjects with scores from -3.00 to +2.80 where a higher score indicates a worse outcome.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Bascom Palmer Eye Institute, Miami, Florida
  - Oregon Health Sciences University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No